CLINICAL TRIAL: NCT07062549
Title: First-in-Human Study of 111In-XYIMSR-01 SPECT/CT in Patients With Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: Study of 111In-XYIMSR-01 SPECT/CT in Patients With Metastatic Clear Cell Renal Cell
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: J20116; IRB00237314 (Other: Johns Hopkins University IRB)
Record Dates: First submitted 2025-06-25; First posted 2025-07-14 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Renal Cell Carcinoma (Kidney Cancer)
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- A (111In-XYIMSR-01) (Experimental): Participants who receive 111In-XYIMSR-01 dosing and SPECT/CT imaging
  Interventions: Drug: 111In-XYIMSR-01

INTERVENTIONS:
Drug: 111In-XYIMSR-01 — Unite Dose: 10.5±1 mCi of 111In-XYIMSR-01 Route of administration: Intravenous catheter placed in an antecubital vein or an equivalent venous access

SUMMARY:
This study is being done to determine if the investigational radiotracer called 111In-XYIMSR-01 is helpful in detecting clear cell renal cell carcinoma tissue in your body when used during a SPECT-CT Scan

ELIGIBILITY:
Inclusion Criteria:

* Males or female sex
* ≥18 years of age
* Willingness to provide signed informed consent and comply with all protocol requirements
* Histological confirmation of RCC with a clear cell component
* 2-10 sites of disease measuring ≥1.5 cm on contrast-enhanced CT and/or MRI imaging of the chest, abdomen and pelvis performed ≤60 days prior to the date of study enrollment
* Screening clinical laboratory values as specified below:

  * Serum bilirubin ≤ 1.5 times the upper limit of normal; for patients with known Gilbert's syndrome, ≤ 3 × ULN is permitted
  * ALT ≤ 3 times the upper limits of normal
  * AST ≤ 3 times the upper limits of normal
  * Creatinine clearance ≥50 mL/min based on Cockcroft-Gault formula
  * Absolute neutrophil count ≥ 1,500 /mm3
  * Platelets ≥100,000/ mm3
  * Hemoglobin ≥ 9.0 g/dL
  * White blood cell count ≥ 2,000/ mm3

Exclusion Criteria:

* Systemic therapy for the treatment of ccRCC within 12 months of study enrollment.
* Subjects administered any radioisotope within five physical half-lives prior to study drug injection.
* Subjects with any medical condition or other circumstances that, in the opinion of the investigator, compromise obtaining reliable data, achieving study objectives, or completion.
* Women of child-bearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the imaging day.
* Women must not be breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | From enrollment to the end of treatment at 1 week
  To evaluate the safety, tolerability, and feasibility of SPECT/CT imaging with 111In-XYIMSR-01 measured by all adverse events according to CTCAE version 5.

SECONDARY OUTCOMES:
Biodistribution assessed by SPECT/CT images | From enrollment to the end of treatment at 1 week
  To determine the biodistribution and radiation dosimetry of 111In-XYIMSR-01
Radiation Dosimetry assessed by SPECT/CT images | From enrollment to the end of treatment at 1 week
  To determine radiation dosimetry of 111In-XYIMSR-01
Total Radioactivity Concentration of 111In-XYIMSR-01 in Plasma Over Time | From enrollment to the end of treatment at 1 week
  To quantify the total radioactivity (expressed in counts per minute [CPM]) in plasma samples at specified time points following injection of 111In-XYIMSR-01
Number of lesions detected | From enrollment to the end of treatment at 1 week
  Investigating the role of 111In-XYIMSR-01 SPECT/CT as a diagnostic assessment tool in comparison to conventional imaging. To compare the number of lesions detected with 111In-XYIMSR-01 SPECT/CT in comparison to conventional imaging all imaging modalities

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Ged, MBBS, Principal Investigator — Johns Hopkins University SKCCC
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States